CLINICAL TRIAL: NCT02815943
Title: Postprandial Metabolism After Bariatric Surgery in Type 2 Diabetes
Acronym: CB4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenured professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-901, 14-176
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Biliopancreatic Diversion; Magnetic Resonance Spectroscopy; Calorimetry, Indirect

ARMS (4):
- Before DBP-DS surgery (Other)
  Interventions: Other: liquid meal; Radiation: PET/scan; Other: [7,7,8,8-2H]-palmitate; Device: indirect calorimetry
- After DBP-DS surgery (Experimental): It is a bariatric surgery. BPD consists in the exclusion of the duodenum from the alimentary tract with re-anastomosis of the blind loop 100 to 150 cm proximal to the ileo-coecal valve. This leads to bypass of the biliopancreatic secretions towards the distal small intestine, resulting in fat malabsorption. BPD also entails a distal gastrectomy to avoid the occurrence of peptic ulceration of the gastrointestinal anastomosis.
  Interventions: Procedure: biliopancreatic diversion with duodenal switch; Other: liquid meal; Radiation: PET/scan; Other: [7,7,8,8-2H]-palmitate; Device: indirect calorimetry
- Before SG surgery (Other)
  Interventions: Other: liquid meal; Radiation: PET/scan; Other: [7,7,8,8-2H]-palmitate; Device: indirect calorimetry
- After SG surgery (Experimental): It is a bariatric surgery where the stomach is reduced to about 15% of its original size, by surgical removal of a large portion of the stomach along the greater curvature.
  Interventions: Procedure: sleeve gastrectomy; Other: liquid meal; Radiation: PET/scan; Other: [7,7,8,8-2H]-palmitate; Device: indirect calorimetry

INTERVENTIONS:
Procedure: biliopancreatic diversion with duodenal switch
  Arms: After DBP-DS surgery
Procedure: sleeve gastrectomy
  Arms: After SG surgery
Other: liquid meal — will be consumed over 30 minutes with [U-13C]-palmitate (0.2 g mixed in the liquid meal) and H2-glucose
Radiation: PET/scan — a dynamic and whole body PET acquisition will be performed on a thoraco-abdominal segment, 150 minutes after an oral administration of 18FTHA
Other: [7,7,8,8-2H]-palmitate — i.v. administration of [7,7,8,8-2H]-palmitate (in 25% human albumin) from time -60 to 360 min.
Device: indirect calorimetry — will be performed every hour throughout the protocol along with exhaled breath collection

SUMMARY:
Bariatric surgery procedures have now been firmly demonstrated to lead to significant improvement and even, in many cases, complete reversal of abnormal glucose homeostasis in type 2 diabetes (T2D). Various surgery procedures are can be performed to induce weight loss. The most striking anti-diabetic effects are observed with biliopancreatic diversion with duodenal switch (BPD-DS), followed by Roux-in-Y gastric bypass (RYGB) and sleeve gastrectomy (SG). The first two procedures induce both a restriction of energy intake and a low absorption of dietary fatty acids while the latter exclusively targets energy intake restriction. The investigator and others have shown that improvement of T2D occurs within days after BPD-DS or RYGB in the vast majority of patients, prior to any significant weight loss. This very rapid metabolic recovery is explained by a normalization of β-cell function after meal challenges and ameliorated hepatic insulin sensitivity. The investigator and others have shown that these acute anti-diabetic effects are mostly recapitulated by matched caloric restriction, independent of changes in gastrointestinal hormones, showing the importance of gastrointestinal-derived energy fluxes for acute diabetes control. Muscle insulin sensitivity, on the other hand, improves more slowly in association with weight loss, demonstrating the heterogeneous metabolic response of the various organs to BPD-DS. Some preliminary studies also demonstrate a rapid reduction of NEFA levels and production rate upon i.v. administration of lipids during euglycemic hyperinsulinemic clamps. This very rapid improvement in NEFA tolerance strongly suggests that adipose tissue storage of circulating fatty acids also improves very rapidly, prior to any significant weight loss, after BPD-DS. It may also suggest an acceleration of oxidative fatty acid metabolism in organs such as the liver, the heart and/or skeletal muscles. Studies of the rapid metabolic changes after bariatric surgery conducted thus far rapidly improved the understanding of the fundamental pathogenic defects of T2D. However, much remains to be understood about the acute changes in gastrointestinal-derived metabolic fluxes, organ-specific metabolic responses to bariatric surgery and their relationship with the reversal of T2D. Using in vivo methodological approaches, the investigator proposes to investigate the early organ-specific changes in dietary fatty acid metabolism in response to BPD-DS vs. SG and their relation to improved systemic changes in glucose homeostasis, insulin sensitivity and β-cell function in patients with T2D.

DETAILED DESCRIPTION:
Participants will undergo a metabolic study before and 8 to 12 days after bariatric surgery after a 12-hour fast and a three-day food and physical activity diary with accelerometry. The patients recover very rapidly from the surgery and will be able to participate to the proposed investigations the week after their hospitalization on an outpatient basis on the earliest week day between 8 and 12 days after the surgery procedure. The metabolic study is a 6-hour meal test using Positron Emitting Tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

Four groups of 11 subjects each: obese subjects with T2D or with normal glucose tolerance undergoing either BPD-DS or SG for treatment of obesity. T2D and control subjects will be matched for age (± 3 years), BMI (± 2 kg/m2) and gender across both BPD-DS and SG.

Exclusion Criteria:

* presence of overt cardiovascular disease, as assessed by history, physical exam, and abnormal EKG;
* treatment with a fibrate, a thiazolidinedione, a beta-blocker or other drugs known to affect lipid or carbohydrate metabolism (except statins, sulfonylurea, metformin, and other antihypertensive agents that can be temporarily stopped prior to the protocols);
* presence of liver or renal disease, uncontrolled thyroid disorder or other major illnesses;
* smoking (>1 cigarette/day) and/or consumption of more than 2 alcoholic beverages per day;
* prior history or current fasting plasma cholesterol level > 7 mmol/l or fasting TG > 6 mmol/l;
* any other contraindication to temporarily stop current medications for hyperglycemia, lipids, or hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
glucose metabolism | 2 years
  will be determined using tracers of glucose
dietary fatty acid uptake | 2 years
  assessed using PET/CT method with oral administration of 18FTHA
whole body inter-organ partitioning | 2 years
  assessed using PET/CT method with oral administration of 18FTHA
lipid metabolism | 2 years
  will be determined using tracers of fatty acids

SECONDARY OUTCOMES:
Dietary fatty acid oxidation rate | 2 years
  will be measured using breath 13CO2 enrichment
Total oxidation rate | 2 years
  will be determined by indirect calorimetry
Hormonal responses | 2 years
  will be determined using a multiplex assay system.
Insulin sensitivity | 2 years
  will be determined using different standard methods, including the HOMA-IR
Insulin secretion index (ISI) | 2 years
  will be assessed using deconvolution of plasma C-peptide with standard C-peptide kinetic parameters
habitual food intake | 2 years
  with a 3-day food record,
physical activity | 2 years
  with portable arm band accelerometry for 3 days prior to each metabolic study

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Carreau AM, Noll C, Blondin DP, Frisch F, Nadeau M, Pelletier M, Phoenix S, Cunnane SC, Guerin B, Turcotte EE, Lebel S, Biertho L, Tchernof A, Carpentier AC. Bariatric Surgery Rapidly Decreases Cardiac Dietary Fatty Acid Partitioning and Hepatic Insulin Resistance Through Increased Intra-abdominal Adipose Tissue Storage and Reduced Spillover in Type 2 Diabetes. Diabetes. 2020 Apr;69(4):567-577. doi: 10.2337/db19-0773. Epub 2020 Jan 8. PMID 31915151